CLINICAL TRIAL: NCT00006565
Title: Randomized Trial to Reduce Environmental Tobacco Smoke in Children With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Bruce P. Lanphear, MD, MPH, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 136; R01HL065731 (NIH)
Record Dates: First submitted 2000-12-01; First posted 2000-12-01 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-10

CONDITIONS: Asthma; Lung Diseases
Keywords: asthma; HEPA; ETS
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HEPA Air Cleaners
  Interventions: Device: HEPA Air Cleaner
- 2 (Placebo Comparator): Inactive (placebo) filtration unit
  Interventions: Device: Placebo Filtration Unit

INTERVENTIONS:
Device: HEPA Air Cleaner — Placement of two active HEPA air cleaners in the homes of children
  Other Names: Austin Healthmate HEPA air cleaner
  Arms: 1
Device: Placebo Filtration Unit — Placement of inactive filtration unit in the homes
  Arms: 2

SUMMARY:
The purpose of this study is to test the effects of reducing indoor environmental tobacco smoke (ETS) on unscheduled asthma visits, asthma symptoms, airway inflammation, and exposure to tobacco smoke measured using air nicotine dosimeters, serum and hair cotinine.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma, a disease characterized by increased airway reactivity and inflammation in response to a variety of stimuli, is emerging as the most prevalent and serious environmental health problem among children in the United States. Numerous studies, both prospective and cross-sectional, suggest that exposure to ETS is one of the predominate risk factors for childhood asthma, but this has not been confirmed in a controlled trial.

DESIGN NARRATIVE:

The randomized, double-blind prospective trial involving 225 children with doctor-diagnosed asthma who are exposed to environmental tobacco smoke tests the efficacy of reducing such exposure on unscheduled asthma visits and asthma symptoms. The intervention consists of placement of 2 high efficiency air filtration with activated carbon, potassium permanganate and zeolite filter insert to reduce exposure to ETS in the experimental homes and inactive (placebo) units in the control group homes. The following hypotheses are tested. (1.0) Children assigned to the ETS reduction group will have a greater than 20 percent reduction in unscheduled asthma visits during one-year follow-up compared with those in the control group. (1.1) Children assigned to the ETS reduction group will have significant improvements in asthma symptoms compared with children in the control group. (1.2) Children assigned to the ETS reduction group will have greater than 10 percent reduction in ETS exposure and exhaled nitric oxide, a measure of airway inflammation during one year of follow-up compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years at enrollment
* Doctor diagnosed asthma by ICD-9 billing codes (from billing records)
* Greater than 1 exacerbation(s) in the past year requiring an unscheduled asthma visit
* Exposed to the smoke of greater than or equal to 5 cigarettes in and around the house per day
* Lived within a 9-county area surrounding the city of Cincinnati

Exclusion Criteria:

* Already using a HEPA air cleaner
* Lacked electricity
* Had a coexisting medical problem
* Family planned to move in the next year

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2000-09; Primary Completion 2003-03 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Unscheduled asthma visits | Measured at 12 months

SECONDARY OUTCOMES:
Asthma symptoms | Measured at 12 months
Exhaled nitric oxide | Measured at 12 months
Tobacco smoke exposure, measured using air nicotine dosimeters, serum cotinine and hair cotinine | Measured at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce P Lanphear, MD, MPH, Principal Investigator — Simon Fraser University

REFERENCES:
- [Result] Wilson SE, Kahn RS, Khoury J, Lanphear BP. Racial differences in exposure to environmental tobacco smoke among children. Environ Health Perspect. 2005 Mar;113(3):362-7. doi: 10.1289/ehp.7379. PMID 15743729
- [Result] Spanier AJ, Hornung RW, Kahn RS, Lierl MB, Lanphear BP. Seasonal variation and environmental predictors of exhaled nitric oxide in children with asthma. Pediatr Pulmonol. 2008 Jun;43(6):576-83. doi: 10.1002/ppul.20816. PMID 18429012
- [Result] Spanier AJ, Hornung R, Lierl M, Lanphear BP. Environmental exposures and exhaled nitric oxide in children with asthma. J Pediatr. 2006 Aug;149(2):220-6. doi: 10.1016/j.jpeds.2006.04.001. PMID 16887438
- [Result] Wilson SE, Kahn RS, Khoury J, Lanphear BP. The role of air nicotine in explaining racial differences in cotinine among tobacco-exposed children. Chest. 2007 Mar;131(3):856-862. doi: 10.1378/chest.06-2123. PMID 17356104
- [Derived] Lanphear BP, Hornung RW, Khoury J, Yolton K, Lierl M, Kalkbrenner A. Effects of HEPA air cleaners on unscheduled asthma visits and asthma symptoms for children exposed to secondhand tobacco smoke. Pediatrics. 2011 Jan;127(1):93-101. doi: 10.1542/peds.2009-2312. Epub 2010 Dec 13. PMID 21149427